CLINICAL TRIAL: NCT04307173
Title: A Phase I Randomised Double-Blind Placebo-Controlled Study of Multiple Ascending Dose of KBL693 in Healthy Participants
Brief Title: Study of Multiple Ascending Dose of KBL693 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: KoBioLabs (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KBL-CURE-2020-01
Record Dates: First submitted 2020-02-21; First posted 2020-03-13 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Moderate to Severe Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): 9 subjects for MAD 1 cohort. 6 subjects on KBL693, 3 subjects on placebo.
  Interventions: Drug: KBL693
- Cohort 2 (Experimental): 9 subjects for MAD 2 cohort. 6 subjects on KBL693, 3 subjects on placebo.
  Interventions: Drug: KBL693

INTERVENTIONS:
Drug: KBL693 — Part 1: 680 mg/day of KBL693 or Placebo;
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort 1
Drug: KBL693 — Part 2: 6800 mg/day of KBL693 or Placebo;
  Route of Administration: Oral
  Other Names: Placebo
  Arms: Cohort 2

SUMMARY:
The study is designed to investigate the safety and tolerability of KBL693 in healthy volunteers. KBL693 has been developed as a potential new treatment for moderate to severe asthma..

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, single centre Phase I study.

Eighteen (18) subjects are planned to be randomised at 1 site across the 2 parts of the study as follows:

* Cohort 1: 680 mg/day
* Cohort 2: 6800 mg/day

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers (also referred to as participants) who can read and understand, and are willing to sign the informed consent form
2. Willing and able to comply with clinic visits (including confinement to CTU) and study-related procedures
3. Male or female healthy volunteers aged ≥18 and ≤65 years at Screening
4. Body mass index (BMI) of ≥18.0 kg/m2 to ≤32 kg/m2 (both inclusive) at Screening
5. Normal hemodynamic parameters: systolic blood pressure (BP) ≥90 mmHg and ≤140 mmHg; diastolic BP ≥50 mmHg and ≤90 mmHg; heart rate (HR) ≥40 bpm and ≤100 bpm at Screening and Day -1. Measurements may be repeated up to 3 times at the discretion of the investigator.

   Please note: participants with out of range values, which are not clinically significant as per the principal investigator's (PI) discretion, will be allowed. The PI may delegate this responsibility to a suitably qualified and trained study team member.
6. The participant is, in the opinion of the PI (or delegate), generally healthy based on assessment of medical history, physical examination, vital signs, ECG, and the results of the haematology, clinical chemistry, urinalysis, serology, and other relevant laboratory tests
7. Baseline laboratory test values within reference ranges based on the blood and urine samples taken at Screening and on Day -1. Out of normal ranges values may be accepted by the PI, if not clinically significant
8. Have regular bowel movements (e.g., once daily)
9. Male participants must agree to practise true abstinence; be surgically sterilised (performed at least 6 months prior); or agree to use of a condom if sexually active with a female partner of childbearing potential, from Screening through 90 days after the final dose of the investigational product (IP).
10. Women of child-bearing potential must agree to practise true abstinence or agree to use effective contraception from Screening through 90 days after the final dose of the IP.

    Effective contraception includes:
    1. Oral contraceptives ("the pill") for at least 1 month prior to Day 1, plus use of a condom
    2. Depot or injectable birth control or implantable contraception (e.g., Implanon) plus use of a condom
    3. Intrauterine device plus use of a condom
    4. Vasectomised male partner (performed at least 6 months prior) who has been documented to no longer produce sperm
11. Women of non-child-bearing potential:

    1. Must have documented evidence of surgical sterilization at least 6 months prior to Screening visit e.g., tubal ligation, hysterectomy.
    2. Must be post-menopausal for at least 12 months prior to Screening, as documented by measurement of follicle stimulating hormone level (≥40 mIU/mL).

Exclusion Criteria:

1. Female participants who are pregnant or lactating
2. The participant's corrected QT interval (QTcF) (Fridericia's correction) is >450 msec (males), and >470 msec (females) at Screening or on Day -1. An out-of-range or abnormal ECG will be repeated at PI's discretion. In total, 3 ECGs should be recorded consecutively at Screening and on Day -1, and the PI (or delegate) must evaluate the triplicate ECG. If the participant's QTcF is >450 msec (males) or >470 msec (females) on at least 2 ECGs or have structural cardiac abnormalities, the participant must be excluded
3. The participant has taken prescription (including antibiotics) or non-prescription medication, herbal remedies, vitamins or minerals, any probiotic drinks and yeast supplements (e.g. Mutaflor®, Bioflor®) within 14 days prior to the first dose of study product unless in the opinion of the PI the medication will not compromise participant safety or interfere with study procedures or data validity. Participant may be rescreened after a washout period of 14 days. Please note use of oral contraceptives and paracetamol up to 2 g/day and/or nonsteroidal anti-inflammatory drugs for symptomatic relief of minor symptoms are allowed
4. Participant has functional GI disorders
5. Participant is a current smoker or has used nicotine containing products within 6 months prior to Screening visit
6. The participant has a substance abuse-related disorder or has a history of drug, alcohol and/or substance abuse deemed significant by the PI
7. The participant has taken any IP within 30 days prior to the first dose of study product or 5 half-lives, whichever is longer
8. The participant has a history of significant hypersensitivity or anaphylaxis involving any drug (including ampicillin, clindamycin or imipenem), any constituent of the IP, food or other precipitating agent (e.g. bee sting). Please note participants with clinically stable mild allergic conditions such as hay fever and mild eczema may be enrolled at the discretion of the PI
9. Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C virus antibody (anti-HCV)at Screening visit.
10. Positive screen for drugs of abuse and cotinine at Screening or on Day -1. Positive screen for alcohol on Day -1.
11. The participant is, in the opinion of the PI, unlikely to comply with the clinical study protocol or is unsuitable for any other reason.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-08-14 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability measure through Adverse Events/Serious Adverse Events | Measurements at Baseline till 28 days
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- blood pressure | Measurement at Baseline till 28 days
  Measured by result of the Vital Sign- blood pressure
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign-heart rate | Measurement at Baseline till 28 days
  Measured by result of the Vital Sign- heart rate
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- axillary body temperature | Measurement at Baseline till 28 days
  Measured by result of the Vital Sign- axillary body temperature
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Vital Sign- respiratory rate | Measurement at Baseline till 28 days
  Measured by result of the Vital Sign- respiratory rate
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through 12-lead ECG | Measurement at Baseline till 28 days
  Measured by result of the ECG measurements and findings
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Physical exam | Measurement at Baseline till 28 days
  Measured by result of the physical exam which includes general appearance, skin, eyes/ears/nose/throat, head and neck, cardiovascular, respiratory, abdomen, extremities, lymph nodes, musculoskeletal and neurologic
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Routine Stool Examination | Measurement at Baseline till 28 days
  Measured by result of the Bristol Stool Examination, Occult blood, Parasites
Safety and tolerability(Incidence of Treatment-Emergent Adverse Events) measure through Clinical laboratory results | Measurement at Baseline till 28 days
  Measured by clinically significant change from baseline clinical laboratory results

SECONDARY OUTCOMES:
Difference in the change from baseline in profile of faecal KBL693 between treatment arms | Measurements at Baseline till 28 days
  Measured by quantitative analysis method for understanding distribution and excretion of KBL693

CONTACTS AND LOCATIONS:
Overall Officials: Lara Hatchuel, Dr, Principal Investigator — Linear Clinical Research
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No